CLINICAL TRIAL: NCT03941379
Title: A Registry of Subjects With Primary Indeterminate Lesions or Choroidal Melanoma
Status: Recruiting | Type: Observational
Sponsor: Aura Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: Registry AU-011-401
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Choroidal Melanoma; Indeterminate Lesions of Eye
Keywords: Choroidal Melanoma; Indeterminate Lesions of Eye
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects previously participated in an Aura Biosciences bel-sar study: Subjects with Choroidal Melanoma or Indeterminate Lesions.

SUMMARY:
The purpose of this observational research study is to follow participants who have been treated with either bel-sar or received alternate treatment (sham, standard of care therapy, etc.) while participating in a previous Aura Biosciences clinical research study to assess the long-term safety and effectiveness in these subjects. This study will collect information from procedures conducted as part of routine follow-up eye care and cancer care. Additionally, the registry will collect all adverse events, information about pregnancy and symptomatic overdose.

DETAILED DESCRIPTION:
This is a multi-center long-term observational Registry of subjects with Primary Indeterminate Lesions or Choroidal Melanoma.

The Registry will initially be open to subjects who have previously participated in an Aura Biosciences bel-sar sponsored clinical trial for their primary Choroidal Melanoma or Indeterminate Lesions.

All subjects will be followed for a minimum of 5 years (including time enrolled in an Aura sponsored clinical trial), until withdrawal of consent, or until death whichever comes first.

No interventions will be required as part of the Registry. Data collection will be based on IL or CM information anticipated to be available based on the standard of care for subjects with CM or IL.

ELIGIBILITY:
Inclusion Criteria:

* Have been clinically diagnosed with primary IL or CM at the time of entry to a previous Aura Biosciences sponsored clinical trial.
* Have received AU-011 bel-sar or assigned to a different cohort or treatment arm (sham, SoC, etc.) an observation cohort in a previous Aura sponsored clinical trial.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with primary Indeterminate Lesions or Choroidal Melanoma who participated in previous Aura Biosciences sponsored clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events and Serious Adverse Events that are related to IL/CM treatment with bel-sar, sham, SoC or alternative treatment. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Aura Biosciences Inc.
Locations (16):
- United States (16):
  - Retina Associates SW, P.C., Tucson, Arizona
  - UCLA Jules Stein Eye Institute, Los Angeles, California
  - Byers Eye Institute at Stanford University, Palo Alto, California
  - Retina Consultants of Sacramento, Sacramento, California
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - W. K. Kellogg Eye Center, University of Michigan, Ann Arbor, Michigan
  - Associated Retinal Consultants, PC, Royal Oak, Michigan
  - Retina Center, Minneapolis, Minnesota
  - Columbia University Medical Center, New York, New York
  - Oregon Health & Science University Casey Eye Institute, Portland, Oregon
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Retina Consultants of Carolina, PA, Greenville, South Carolina
  - St. Thomas Health / Tennessee Retina, PC, Nashville, Tennessee
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Houston, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ocular Melanoma — http://www.ocularmelanoma.org/